CLINICAL TRIAL: NCT01755195
Title: A Phase 2 Study of Cabozantinib (XL184), a Dual Inhibitor of MET and VEGFR, in Patients With Metastatic Refractory Soft Tissue Sarcoma
Brief Title: Cabozantinib for Adults With Advanced Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alice Chen, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130044; 13-C-0044
Record Dates: First submitted 2012-12-18; First posted 2012-12-24 (Estimated); Results first posted 2021-09-16 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Refractory Soft Tissue Sarcomas
Keywords: Dual Inhibitor of MET and VEGFR; XL184; Metastatic Refractory; Soft Tissue Sarcoma; Rare Heterogeneous Tumor
MeSH Terms: conditions — Sarcoma | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cabozantinib (Experimental): 60 mg tablets orally once a day in a 28-day cycle.
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib inhibits multiple receptor tyrosine kinases (RTKs) implicated in tumor growth, metastasis, and angiogenesis, and targets primarily mesenchymal-epithelial transition factor (MET) and vascular endothelial growth factor receptor 2 (VEGFR2).
  Other Names: Cometriq

SUMMARY:
Background:

- Cabozantinib is a cancer treatment drug that blocks the growth of new blood vessels in tumors. It can also block a chemical on tumor cells that allows the cells to grow. A similar drug, pazopanib, is used to treat types of cancer known as sarcomas. Researchers want to see if cabozantinib can be an effective treatment for types of soft tissue sarcoma that have not responded to earlier treatments.

Objectives:

- To test the effectiveness of cabozantinib for soft tissue sarcomas that have not responded to standard treatments.

Eligibility:

- Individuals at least 18 years of age who have soft tissue sarcomas that have not responded to standard treatments.

Design:

* Participants will be screened with a physical exam and medical history. Blood samples will be collected. Imaging studies and other tests will be used to study the tumor before the start of treatment.
* Participants will take cabozantinib tablets daily for 28-day cycles of treatment. The tablets should be taken whole on an empty stomach.
* Treatment will be monitored with frequent blood tests and imaging studies.
* Participants will continue to take cabozantinib for as long as the tumor does not become worse and the side effects are not too severe.

DETAILED DESCRIPTION:
Background:

* Soft tissue sarcomas (STS) are a relatively rare heterogeneous group of tumors that constitute about 1% of adult cancers.
* The mainstay of treatment for advanced disease has been palliative chemotherapy with a median overall survival of approximately 12 months. This has not changed considerably in the past years and there is an unmet need for newer targeted therapies.
* Vascular endothelial growth factor (VEGF) levels are elevated in patients with STS and various sarcoma cell lines express high levels of activated c-Met receptor.
* We hypothesize that dual targeting of the VEGF and mesenchymal-epithelial transition factor (c-MET) pathways with cabozantinib would result in clinical benefit in patients with soft tissue sarcoma.

Objectives:

Primary:

* Assess the response rate (Complete Response (CR)+Partial Response (PR) of cabozantinib in patients with soft tissue sarcomas.
* Assess the 6 month progression free survival (PFS) of cabozantinib in soft tissue sarcomas.

Secondary:

-Determine and compare circulating levels of hepatocyte growth factor (HGF), soluble MET (sMET), VEGF-A, and soluble vascular endothelial growth factor receptor 2 (VEGFR2) (sVEGFR2) prior to and following administration of cabozantinib.

Eligibility:

* Patients must have had disease progression following one line of standard therapy
* Age greater than or equal to 18 years.
* Adequate organ function.

Design:

* All patients will receive cabozantinib at 60 mg by mouth (PO) daily in 4 week cycles.
* Tumor response evaluations by imaging will be done every 2 cycles (less frequently for patients on study more than one year).
* The study will be conducted as a dual-endpoint two-stage Phase II trial to target objective tumor response rate (CR+PR) of 30% against an unacceptably low rate of 10%, and 6-month PFS rate of 65% against an unacceptably low rate of 45% (corresponding to median PFS of 9.6 vs. 5.2 months).
* The trial will accrue up to 55 patients.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically or cytologically confirmed soft tissue sarcoma that is metastatic or unresectable and for which standard treatment that prolongs survival does not exist or is no longer effective.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >20 mm with conventional techniques or as >10 mm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam.
* Patients are allowed prior vascular endothelial growth factor receptor (VEGFR)-tyrosine kinase inhibitors (TKI) therapy.
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of cabozantinib in patients <18 years of age, children are excluded from this study.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 1 (Karnofsky >70%).
* Life expectancy > 3 months.
* Patients must have normal organ and marrow function as defined below:

  * leukocytes greater than or equal to 3,000/mcL
  * absolute neutrophil count greater than or equal to 1,500/mcL
  * platelets greater than or equal to 100,000/mcL
  * total bilirubin less than or equal to 1.5 times ULN
  * Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase(SGOT)/alanine aminotransferase (ALT) serum glutamic pyruvic transaminase(SGPT) less than or equal to 2.5 times institutional upper limit of normal creatinine within normal institutional limits
  * creatinine within normal institutional limits OR clearance greater than or equal to 60 mL/min/1.73 m(2) for patients with creatinine levels above institutional normal.
  * hemoglobin greater than or equal to 9 g/dL
  * serum albumin greater than or equal to 2.8g/dL
  * lipase <2.0 times upper limit of normal (ULN) and no radiologic or clinical evidence of pancreatitis
  * urine protein/creatinine ratio (UPCR) less than or equal to 1
  * serum phosphorus calcium, magnesium and potassium greater than or equal to lower limit of normal (LLN)
* Subjects must have blood pressure (BP) no greater than 140 mmHg (systolic) and 90 mmHg (diastolic) for eligibility. Initiation or adjustment of BP medication is permitted prior to study entry provided that the average of three BP readings at the time of enrollment is less than or equal to 140/90 mmHg
* Patients must be able to swallow whole tablets. Tablets must not be crushed or chewed.
* The effects of cabozantinib on the developing human fetus are unknown. For this reason and because receptor tyrosine kinases are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception. All subjects of reproductive potential must agree to use both a barrier method and a second method of birth control during the course of the study and for 4 months after the last dose of study drug(s).

Sexually active subjects (men and women) must agree to use medically accepted barrier methods of contraception (e.g., male or female condom) during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used.

-Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients who have had anticancer therapy, including kinase inhibitors or any investigational agent within 4 weeks or 5 half-lives (whichever is shorter) (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered to baseline from adverse events (except alopecia and other non-clinically significant adverse events (AEs). Patients who have received prior cabozantinib or inhibitors of tyrosine-protein kinase mesenchymal epithelial transition factor (c-MET) or hepatocyte growth factor (HGF) are ineligible.
* The subject has received radionuclide treatment within 6 weeks of the first dose of study treatment
* The subject has received radiation therapy within 4 weeks (greater than or equal to 2 weeks for palliative radiation therapy)
* Patients with active brain metastases or carcinomatous meningitis or epidural disease are excluded from this clinical trial. Subjects with brain metastases previously treated with whole brain radiation or radiosurgery or subjects with epidural disease previously treated with radiation who are asymptomatic and have remained stable for 4 weeks and do not require steroid treatment for at least 2 weeks before starting study treatment are eligible. Neurosurgical resection of brain metastases or brain biopsy is permitted if completed at least 3 months before starting study treatment. Baseline brain imaging with contrast-enhanced CT or MRI scans for subjects with known brain metastases is required to confirm eligibility.
* Eligibility of subjects receiving any medications or substances known to affect or with the potential to affect the activity of cabozantinib will be determined following review of their cases by the Principal Investigator. Patients who are taking enzyme-inducing anticonvulsant agents are not eligible.
* Patients with refractory nausea and vomiting, chronic gastrointestinal diseases (e.g., inflammatory bowel disease), or significant bowel resection that could interfere with absorption.
* Uncontrolled intercurrent illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because cabozantinib has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with cabozantinib, breastfeeding should be discontinued if the mother is treated with cabozantinib.
* Strong inhibitors and inducers of cytochrome P450 3A4 (CYP3A4) can affect levels of cabozantinib and should be avoided whenever possible or switched to alternatives. Subjects requiring chronic concomitant treatment of strong CYP3A4 inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentine, phenobarbital, and St. John's Wort) are not eligible for this study. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/; medical reference texts such as the Physicians Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over the-counter medicine or herbal product.
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with cabozantinib. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* The subject requires concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, heparin, thrombin or Factor Xa inhibitors, or antiplatelet agents (e.g., clopidogrel). Low dose aspirin (less than or equal to 81 mg/day), low-dose warfarin (less than or equal to 1 mg/day), and prophylactic low molecular weight heparin (LMWH) are permitted. (Please note that there may be cases in which patients on study require anticoagulation for deep vein thrombosis (DVT)/pulmonary embolism (PE) management; this does not necessitate taking

the patient off study.)

* The subject has experienced any of the following

  * clinically-significant gastrointestinal bleeding within 6 months before the first dose of study treatment
  * hemoptysis of greater than or equal to 0.5 teaspoon (2.5 mL) of red blood within 3 months before the first dose of study treatment
  * any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment
* The subject has radiographic evidence of cavitating pulmonary lesion(s).
* The subject has tumor in contact with, invading, or encasing any major blood vessels
* The subject has evidence of tumor invading the gastrointestinal (GI) tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  1. Cardiovascular disorders including:

     1. Congestive heart failure (CHF): New York Heart Association (NYHA) Class III (moderate) or Class IV (severe) at the time of screening
     2. Concurrent uncontrolled hypertension defined as sustained BP > 140 mm Hg systolic, or > 90 mm Hg diastolic despite optimal antihypertensive treatment within 7 days of the first dose of study treatment
     3. Any history of congenital long QT syndrome
     4. Any of the following within 6 months before the first dose of study treatment:

        * unstable angina pectoris
        * clinically-significant cardiac arrhythmias
        * stroke (including transient ischemic attack (TIA), or other ischemic event)
        * myocardial infarction
        * thromboembolic event requiring therapeutic anticoagulation (Note: subjects with a venous filter (e.g. vena cava filter) are not eligible for this study)
  2. Gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation including:

     1. Any of the following within 28 days before the first dose of study treatment

        * intra-abdominal tumor/metastases invading GI mucosa
        * active peptic ulcer disease,
        * inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis
        * malabsorption syndrome
     2. Any of the following within 6 months before the first dose of study treatment:

        * abdominal fistula
        * gastrointestinal perforation
        * bowel obstruction or gastric outlet obstruction
        * intra-abdominal abscess. Note: Complete resolution of an intra-abdominal abscess must be confirmed prior to initiating treatment with cabozantinib even if the abscess occurred more that 6 months before the first dose of study treatment.
  3. Other disorders associated with a high risk of fistula formation including percutaneous endoscopic gastrostomy (PEG) tube placement within 3 months before the first dose of study therapy
  4. Other clinically significant disorders such as:

     1. serious non-healing wound/ulcer/bone fracture within 28 days before the first dose of study treatment
     2. history of organ transplant, including allogeneic bone marrow transplant
     3. concurrent uncompensated hypothyroidism or thyroid dysfunction within 7 days before the first dose of study treatment
     4. history of major surgery as follows:

     i. Major surgery within 3 months of the first dose of cabozantinib if there were no wound healing complications or within 6 months of the first dose of cabozantinib if there were wound complications

     ii. Minor surgery within 1 months of the first dose of cabozantinib if there were no wound healing complications or within 3 months of the first dose of cabozantinib if there were wound complications

     In addition, complete wound healing from prior surgery must be confirmed at least 28 days before the first dose of cabozantinib irrespective of the time from surgery
* The subject is unable to swallow tablets
* The subject has a corrected QT interval calculated by the Fridericia formula (QTcF) >500 ms within 28 days before enrollment. Note: if initial QTcF is found to be > 500 ms, two additional EKGs separated by at least 3 minutes should be performed. If the average of these three consecutive results for QTcF is less than or equal to 500 ms, the subject meets eligibility in this regard.
* The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.
* The subject has had evidence within 2 years of the start of study treatment of another malignancy which required systemic treatment.
* Patients should not have any clinical evidence of an active infection at the time of enrollment.

INCLUSION OF WOMEN AND MINORITIES:

Both men and women of all races and ethnic groups are eligible for this trial.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-01-15 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2023-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice P Chen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coindre JM, Terrier P, Guillou L, Le Doussal V, Collin F, Ranchere D, Sastre X, Vilain MO, Bonichon F, N'Guyen Bui B. Predictive value of grade for metastasis development in the main histologic types of adult soft tissue sarcomas: a study of 1240 patients from the French Federation of Cancer Centers Sarcoma Group. Cancer. 2001 May 15;91(10):1914-26. doi: 10.1002/1097-0142(20010515)91:103.0.co;2-3. PMID 11346874
- [Background] Edmonson JH, Ryan LM, Blum RH, Brooks JS, Shiraki M, Frytak S, Parkinson DR. Randomized comparison of doxorubicin alone versus ifosfamide plus doxorubicin or mitomycin, doxorubicin, and cisplatin against advanced soft tissue sarcomas. J Clin Oncol. 1993 Jul;11(7):1269-75. doi: 10.1200/JCO.1993.11.7.1269. PMID 8315424
- [Background] Elias A, Ryan L, Sulkes A, Collins J, Aisner J, Antman KH. Response to mesna, doxorubicin, ifosfamide, and dacarbazine in 108 patients with metastatic or unresectable sarcoma and no prior chemotherapy. J Clin Oncol. 1989 Sep;7(9):1208-16. doi: 10.1200/JCO.1989.7.9.1208. PMID 2504890
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-C-0044.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cabozantinib
Started | 55
Completed | 42
Not Completed | 13
Not completed — Participant noncompliance | 2
Not completed — Switched to alternative treatment | 4
Not completed — Withdrawal by Subject | 1
Not completed — Participant refused to start treatment | 1
Not completed — Participant has been consented for another trial | 1
Not completed — Refused further treatment | 3
Not completed — Complicating disease/intercurrent illness | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cabozantinib
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.69 (12.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 33
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (Complete Response (CR)+Partial Response (PR) of Cabozantinib in Patients With Soft Tissue Sarcomas
Description: Objective response was assessed by the Response Evaluation Criteria in Solid Tumors RECIST) v1.1. Complete Response is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Date treatment consent signed to date off study, approximately 86 months and 3 days.
Population: 1/55 participants did not start therapy.
Measure: Number (95% Confidence Interval); unit: percentage of particpants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 54
percentage of particpants | 11.1 [4.2 to 22.6]

2. Primary Outcome: Percentage of Participants With 6 Month Progression Free Survival (PFS)
Description: Progression in participants with soft tissue sarcomas treated with cabozantinib was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Progression is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The appearance of one or more new lesions is also considered progressions.
Time Frame: 6 months
Population: 1/55 participants did not start therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 54
percentage of participants | 49.3 [36.2 to 67.3]

3. Secondary Outcome: Mean Change From Baseline in Levels of Circulating Hepatocyte Growth Factor (HGF)
Description: Blood samples were collected before treatment on the first day of cycles 1 and 2 to determine circulating levels of HGF. HGF protein content (in picograms; pg) in blood plasma (in milliliters; mL) was measured for each sample with a two-site immunoassay and the difference from before to after treatment for each patient was reported. A change in this biomarker from the baseline value has not been linked to clinical outcomes; that is, it is neither a good or a bad outcome.
Time Frame: Baseline to Cycle 1 Day 1 and baseline to Cycle 2 Day 1
Population: 42/54 participants were analyzed for this outcome measure. One participant did not start therapy, and twelve participants did not participate in the optional biomarker testing.
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Cabozantinib
Number analyzed (Participants) | 42
pg/mL
  Baseline to Cycle 1 Day 1 | -51.3 [-235.5 to 151.0]
  Baseline to Cycle 2 Day 1 | 344.8 [4.1 to 685.6]

4. Secondary Outcome: Mean Change From Baseline in Levels of Circulating Soluble Mesenchymal Epithelial Transition Factor (sMET)
Description: Blood samples were collected before treatment on the first day of cycles 1 and 2 to determine circulating levels of soluble MET (sMET). sMET protein content (in nanograms; ng) in blood plasma (in milliliters; mL) was measured for each sample with a two-site immunoassay and the difference from before to after treatment for each patient was reported. A change in this biomarker from the baseline value has not been linked to clinical outcomes; that is, it is neither a good or a bad outcome.
Time Frame: Baseline to Cycle 1 Day 1 and baseline to Cycle 2 Day 1
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Cabozantinib
Number analyzed (Participants) | 42
ng/mL
  Baseline to Cycle 1 Day 1 | -6.1 [-12.0 to -0.3]
  Baseline to Cycle 2 Day1 | 16.4 [3.4 to 29.4]

5. Secondary Outcome: Mean Change From Baseline in Levels of Circulating Vascular Endothelial Growth Factor A (VEGF-A)
Description: Blood samples were collected before treatment on the first day of cycles 1 and 2 to determine circulating levels of VEGF-A. VEGF-A protein content (in picograms; pg) in blood plasma (in milliliters; mL) was measured for each sample with a two-site immunoassay and the difference from before to after treatment for each patient was reported. A change in this biomarker from the baseline value has not been linked to clinical outcomes; that is, it is neither a good or a bad outcome.
Time Frame: Baseline to Cycle 1 Day 1 and baseline to Cycle 2 Day 1
Population: as for outcome 3
Measure: Mean (97.5% Confidence Interval); unit: pg/mL
Arm/Group | Cabozantinib
Number analyzed (Participants) | 42
pg/mL
  Baseline to Cycle 1 Day 1 | 5.6 [-3.6 to 14.7]
  Baseline to Cycle 2 Day 1 | 32.5 [6.5 to 58.5]

6. Secondary Outcome: Mean Change From Baseline in Levels of Circulating Soluble Vascular Endothelial Growth Factor Receptor 2 (sVEGFR-2)
Description: Blood samples were collected before treatment on the first day of cycles 1 and 2 to determine circulating levels of soluble VEGFR2 (sVEGFR-2). sVEGFR-2 protein content (in nanograms; ng) in blood plasma (in milliliters; mL) was measured for each sample with a two-site immunoassay and the difference from before to after treatment for each patient was reported. A change in this biomarker from the baseline value has not been linked to clinical outcomes; that is, it is neither a good or a bad outcome..
Time Frame: Baseline to Cycle 1 Day 1 and baseline to Cycle 2 Day 1
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Cabozantinib
Number analyzed (Participants) | 42
ng/mL
  Baseline to Cycle 1 Day 1 | -1.0 [-2.6 to 0.6]
  Baseline to Cycle 2 Day 1 | -10.9 [-13.5 to -8.4]

7. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 86 months and 3 days.
Population: 1/55 participants did not start therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib
Number analyzed (Participants) | 54
Participants | 53

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 86 months and 3 days.
Description: 1/55 participants did not start therapy.
Arm/Group | Cabozantinib
All-Cause Mortality (participants affected / at risk) | 3/54
Serious Adverse Events (participants affected / at risk) | 14/54
Other Adverse Events (participants affected / at risk) | 53/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabozantinib (N=54)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
General disorders and administration site conditions - Other, fever (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Serum amylase increased (Investigations) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Stroke (Nervous system disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 3 (4)
Tooth infection (Infections and infestations) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabozantinib (N=54)
Abdominal pain (Gastrointestinal disorders) | 9 (25)
Activated partial thromboplastin time prolonged (Investigations) | 6 (14)
Alanine aminotransferase increased (Investigations) | 29 (59)
Alkaline phosphatase increased (Investigations) | 22 (28)
Allergic reaction (Immune system disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (9)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 13 (32)
Anorexia (Metabolism and nutrition disorders) | 19 (30)
Anxiety (Psychiatric disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 25 (51)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8)
Bladder perforation (Renal and urinary disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (3)
Blood and lymphatic system disorders - Other, Blood in stool due to hemorrhoids (Blood and lymphatic system disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 3 (7)
Blurred vision (Eye disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Brachial plexopathy (Nervous system disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 9 (10)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
CPK increased (Investigations) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 3 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Chills (General disorders) | 5 (5)
Concentration impairment (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 17 (24)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Creatinine increased (Investigations) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 7 (10)
Dental caries (Gastrointestinal disorders) | 1 (2)
Depression (Psychiatric disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 28 (70)
Dizziness (Nervous system disorders) | 12 (17)
Dry eye (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 12 (19)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (10)
Dysgeusia (Nervous system disorders) | 17 (24)
Dyspepsia (Gastrointestinal disorders) | 10 (11)
Dysphagia (Nervous system disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 (15)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 7 (10)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 4 (4)
Endocrine disorders - Other, Lactate dehydrogenase increased (Endocrine disorders) | 1 (1)
Enterocolitis (Infections and infestations) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Eye disorders - Other, Eye disorders; erythrodysesthesia syndrome (Eye disorders) | 1 (1)
Eye disorders - Other, Eye disorders; loss of peripheral vision (Eye disorders) | 1 (2)
Eye disorders - Other, High Spatial Frequencies (Eye disorders) | 1 (1)
Eye disorders - Other, Vision change (black spots) (Eye disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 24 (48)
Fever (General disorders) | 6 (6)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Flashing lights (Eye disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 7 (9)
Flu like symptoms (General disorders) | 5 (5)
Flushing (Vascular disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (5)
Gastrointestinal disorders - Other, GI:Increased Salivation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, Gastrointestinal disorders - Other, specify: Rectal discharge (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, blood in stool (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, intermittent decrease/loss of appetite (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, loose stool (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions - Other, Mouth Sores (General disorders) | 1 (1)
General disorders and administration site conditions - Other, Numbness of Tongue (General disorders) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 2 (2)
Gum infection (Infections and infestations) | 1 (3)
Hair color changes (Skin and subcutaneous tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 20 (45)
Hematuria (Renal and urinary disorders) | 7 (9)
Hemoglobinuria (Renal and urinary disorders) | 4 (5)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 9 (11)
Hot flashes (Metabolism and nutrition disorders) | 5 (5)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (9)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (9)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (4)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 43 (437)
Hyperthyroidism (Endocrine disorders) | 2 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 17 (38)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (13)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (4)
Hypokalemia (Metabolism and nutrition disorders) | 7 (10)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (10)
Hyponatremia (Metabolism and nutrition disorders) | 5 (19)
Hypophosphatemia (Metabolism and nutrition disorders) | 14 (27)
Hypotension (Vascular disorders) | 4 (8)
Hypothyroidism (Endocrine disorders) | 19 (27)
Infections and infestations - Other, Facial infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, Infection - Tumor fungation (Infections and infestations) | 1 (1)
Infections and infestations - Other, Malaria (Infections and infestations) | 1 (1)
Infections and infestations - Other, Post-dental work (Infections and infestations) | 1 (1)
Infections and infestations - Other, Urine (Infections and infestations) | 1 (1)
Infections and infestations - Other, Viral Infection (Infections and infestations) | 1 (1)
Injury, poisoning and procedural complications - Other, Urine PCR (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5)
Investigations - Other, Hyperphosphatemia (Investigations) | 1 (1)
Investigations - Other, Lactate dehydrogenase increased (Investigations) | 1 (1)
Investigations - Other, Protein total decreased (Investigations) | 3 (5)
Investigations - Other, Total protein decreased (Investigations) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 4 (4)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Lipase increased (Investigations) | 11 (24)
Lymphocyte count decreased (Investigations) | 13 (46)
Malaise (General disorders) | 1 (2)
Memory impairment (Nervous system disorders) | 2 (2)
Metabolism and nutrition disorders - Other, Early Satiety (Metabolism and nutrition disorders) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1)
Mucosal infection (Infections and infestations) | 4 (4)
Mucositis oral (Gastrointestinal disorders) | 14 (33)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, intermittent muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (16)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Nail infection (Infections and infestations) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Nausea (Gastrointestinal disorders) | 24 (56)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (9)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — (incl cysts and polyps) - Other, Bleeding from tumor site
Neuralgia (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 13 (71)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 3 (4)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 9 (11)
Pain (General disorders) | 10 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (14)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (3)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 29 (55)
Paresthesia (Nervous system disorders) | 3 (3)
Periodontal disease (Gastrointestinal disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Platelet count decreased (Investigations) | 16 (23)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Presyncope (Nervous system disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 13 (27)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Radiculitis (Nervous system disorders) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4)
Rectal pain (Gastrointestinal disorders) | 2 (2)
Renal and urinary disorders - Other, Dysuria (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) — Nephrotic syndrome: Albumin 2.9 low, 24 hr Urine protein 3.58 , Edema.
Renal and urinary disorders - Other, Protein Creatinine Ratio Increased (Renal and urinary disorders) | 1 (2)
Renal and urinary disorders - Other, Urine protein-Creatinine ratio increased (Renal and urinary disorders) | 2 (2)
Renal and urinary disorders - Other, elevated protein/creatinine ratio (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, hesitancy (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, proteinuria (Renal and urinary disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, URI with cold (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Serum amylase increased (Investigations) | 7 (59)
Sinus bradycardia (Cardiac disorders) | 4 (5)
Sinus tachycardia (Cardiac disorders) | 4 (5)
Sinusitis (Infections and infestations) | 2 (2)
Skin and subcutaneous tissue disorders - Other, B/L lower extremity lacerations; (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Cellulitis with fistula (supra-pubic area-LLQ) (Skin and subcutaneous tissue disorders) | 1 (2)
Skin and subcutaneous tissue disorders - Other, Chest Redness (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Erythema along port (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Graft dehiscence (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Hair hypopigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, Hair thinning (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, Lump on upper L chest wall (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Pruritus /Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Seborrheic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Skin and subcutaneous tissue disorders - Other, specify: Hair color change
Skin and subcutaneous tissue disorders - Other, Skin and subcutaneous tissue disorders - Other: hair (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Skin discoloration (over R shoulder) (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Skin lumps (face, ear, hairline) (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, fingernail splitting (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, hair lightening (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, hand purple/blue discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, intermittent petechiae bilateral breast (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, pin-size hole over port (no drainage) (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, sore on elbow (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, sunburn from swimming; chest, back, BUE (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (3) — Skin and subcutaneous tissue disorders - Other, specify: Hair color change
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 10 (12)
Skin infection (Infections and infestations) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 12 (13)
Spasticity (Nervous system disorders) | 4 (4)
Stomach pain (Gastrointestinal disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 3 (3)
Thyroid stimulating hormone increased (Investigations) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Tooth development disorder (Gastrointestinal disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Toothache (Gastrointestinal disorders) | 4 (4)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (9)
Upper respiratory infection (Infections and infestations) | 7 (10)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (6)
Urinary tract pain (Renal and urinary disorders) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 (2)
Vaginal infection (Infections and infestations) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 17 (41)
Weight loss (Investigations) | 16 (49)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
White blood cell decreased (Investigations) | 19 (71)
weight loss (Investigations) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Endocrine disorders - Other, TSH decreased (Endocrine disorders) | 1 (1)
Soft tissue necrosis lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Surgical and medical procedures - Other, Teeth extractions (Surgical and medical procedures) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/95/NCT01755195/Prot_SAP_002.pdf
  • Informed Consent Form (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/95/NCT01755195/ICF_001.pdf